CLINICAL TRIAL: NCT03011840
Title: Effect of Patient Information Leaflet on Working Pattern and Patient Satisfaction Level in a Busy Indian Day Care Operative Theatre Complex
Brief Title: Effect of Patient Information Leaflet on Working Pattern and Patient Satisfaction Level for Day Care Surgeries.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Sumitra G Bakshi, Professor and Anesthetist, Tata Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Project no 1775
Record Dates: First submitted 2017-01-02; First posted 2017-01-05 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Patient Compliance
Keywords: Patient education handout; Patient satisfaction
MeSH Terms: conditions — Patient Compliance; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre intervention (No Intervention): In the first part planned over 2months (Jan - Feb), feedback forms will be collected from patients at the end of minor OT procedure. The number of postponement or rescheduling of cases will be noted.
  Postponement or rescheduling of case is defined as an event when the patient who is called for his turn in minor OT is deferred for any amount of time in account of starvation not adequate, investigations not brought, medications not taken as prescribed.
- Post Intervention (Experimental): In the intervention phase, the patient information leaflet (PIL) will be handed over to all patients planned for procedure in the minor OT complex. This leaflet will be handed over by the attending doctor in the Head neck OPD. The checklist pertaining to counselling at the Head neck OPD will be ticked after they are carried out. The patient will be instructed to read leaflet carefully and carry the leaflet on the day of Minor OT procedure. In the minor OT the discharge checklist in the PIL would be carried out by all concerned including the surgical, anesthesia and nursing team. The impact of use of PIL will be assessed by noting the number of postponement or rescheduling of cases.
  Interventions: Other: Information leaflet

INTERVENTIONS:
Other: Information leaflet — Patient information leaflet with instructions to be carried out before procedure under general anesthesia
  Arms: Post Intervention

SUMMARY:
This study aims to understand the benefits of imparting pre operative instructions through written leaflets. The influence on the number of avoidable postponements and delay is also studied.The study is restricted to patients undergoing Head & Neck procedures under General Anaesthesia, at the minor OT complex at Tata Memorial Hospital

DETAILED DESCRIPTION:
INTRODUCTION:

Patient Information is one of the key determinants of patient satisfaction. Adequate information about the disease condition, treatment plan, waiting times and 'what to do next' affects patients' overall satisfaction level. Good quality information not only reduces patient anxiety and stress, but also reduces unreasonable expectations and misconceptions. Patient satisfaction has always remained an important and commonly used indicator for measuring the quality in health care.

In the recent years there is a gradual upward trend in day care surgeries all across the globe; an estimated 83% of the surgeries in the United States being performed on an ambulatory basis. In India, about 20 percent of all surgical procedures are performed on outpatients. It is estimated that by 2020, 75 percent of all surgical operations in India will be carried out in ambulatory surgery centers. The increasing trend of ambulatory surgeries has emerged from advances in anesthesia and surgical techniques. Patient information and effective communication is critical in these surgeries especially the ones that need General Anesthesia.

Provision of information is one of the mainstays of effective day surgery management. This needs to cover not only what to do before and after surgery, but also what will happen on the day of surgery. There are several ways of providing information like written information, using a video, over telephone or by patient interviews before and after surgery. Verbal information alone is inadequate and must be reinforced with well-presented printed material.

Tata Memorial Hospital is a premier tertiary level cancer hospital in India. Around 140-150 patients undergo minor surgical procedures (diagnostic and therapeutic) in the Minor OT complex every day. About 30-40% of surgeries belong to the Head & Neck region alone.About 40-50% of these surgeries are done under general anesthesia. At present the communication with patients in the busy outpatient department is mainly verbal. Due to time constrains, lack of a responsible attendant with the patient, important information with respect to the day care procedure is often not effectively delivered. This leads to patients not following instruction adequately with respect to starvation, medications to be taken on the day of the procedure and also not carrying all essential documents. This leads to delays, rescheduling of cases and rarely postponement of procedures.

Does an information leaflet provide an effective way of communication in the peri-procedure period? Will it help in better information delivery and hence reduce the number of avoidable postponements and delay. And does this translate to better patient satisfaction is want this study aims to see. The study is restricted to patients undergoing Head & Neck procedures under general anesthesia, as they form the major bulk of patients in our minor OT complex and for logistic reasons to start with a defined group of patients.

AIMS AND OBJECTIVES:

1. To reduce postponement of cases due to lack of information to patients prior to the procedure.
2. To compare satisfaction levels between patients , before and after introduction of information leaflet

Primary end point:

To reduce postponement of cases due to lack of information to patients prior to the procedure.

Secondary end point To compare satisfaction levels between patients, before and after introduction of information leaflet.

Design of the study: Intervention

MATERIAL AND METHODS

After Institutional Review Board approval, all adult patients meeting inclusion criteria and undergoing surgeries in the Minor operation theater 'OT' complex during a 5 month period will be enrolled in the study. The study will be done in two parts.

In the First half of study- planned over 2 months (Jan - Feb), feedback forms will be collected from patients at the end of minor 'OT' procedure. All patients, meeting inclusion criteria, at the end of the procedure prior to discharge from the minor 'OT' will be explained about the study and they shall be given a feedback form to be filled and submitted. Also the number of postponement or rescheduling of cases will be noted.

Postponement or rescheduling of case is defined as an event when the patient who is called for his turn in minor 'OT' is deferred for any amount of time in account of starvation not adequate, investigations not brought, medications not taken as prescribed.Any postponement in view of awaiting opinion form senior consultant , special equipment or any investigations called in view of patients clinical conditions which was not anticipated in the Out Patient Department 'OPD' by the surgical colleague, or due to lack of OT time will not be included.

After the initial collection of feedback over 2 months, the patient information leaflet (PIL) will be handed over to all patients planned for procedure in the minor 'OT' complex (Second half of study). This leaflet will be handed over by the attending doctor in the Head neck 'OPD'. The checklist pertaining to counselling at the Head neck 'OPD' will be ticked after they are carried out. The patient will be instructed to read leaflet carefully and carry the leaflet on the day of Minor OT procedure. In the minor OT the discharge checklist in the 'PIL' would be carried out by all concerned including the surgical, anesthesia and nursing team. A period of 1 month will be allowed to streamline the use of patient information leaflet.

In the subsequent 2 months,Apr- May , the impact of use of 'PIL' will be assessed. Firstly by noting the number of postponement or rescheduling of cases. In addition all patients meeting inclusion criteria will be given the feedback form. at the end of their procedure in minor 'OT'.

For patients coming to minor 'OT' without a patient information leaflet- one would ascertain if the leaflet was handed in 'OPD' and not brought to minor OT or if the leaflet was not handed at all. The numbers of such misses will be recorded.Patients who did not get the leaflet in the 'OPD' will be excluded from study.

Sample size calculation:

From the investigator's preliminary review of postponement rate at the study center is around 20%. The investigators aim for a reduction in postponement by 50%. Group sample sizes of 199 in group 1 and 199 in group 2 achieve 80.007% power to detect a difference between the group proportions of -0.1000. The proportion in group 1 (the treatment group) is assumed to be 0.2000 under the null hypothesis and 0.1000 under the alternative hypothesis. The proportion in group 2 (the control group) is 0.2000. The test statistic used is the two-sided Z-Test with pooled variance. The significance level of the test is 0.0500.Considering a 20% loss to follow up from 'OPD' to minor 'OT', the sample size needed is 480 patients.On an average at least 250 patients of head neck patients undergo procedure under general anesthesia, per month (12-15 patients /day x 20 working days). With due consideration of our inclusion criteria, a two month recruitment period before and after the intervention should be adequate.

MEASUREMENTS

* No. of cases postponed before and after the introduction of the leaflet and reasons behind them
* Primary data collected will be patient satisfaction levels after the procedure (both pre and post 'PIL') on a 5 point Likert scale (Ranging from very poor = 0 to Excellent = 4)
* No of patients who did not receive the patient information leaflet in the' OPD'
* No of patients who received the Patient information leaflet but did not get it along to the minor OT

STATISTICAL ANALYSIS All Data will be analyzed using Statistical Analysis Software Package (SPSS) software. Likert scores will be treated as ordinal data. Proportions will be compared using chi square analysis. Additionally Multivariate logistic regression analysis will be used to assess the contribution of possible covariates, including age sex and patient knowledge on patient satisfaction. For all data P-value < 0.05 will be considered as statistical significant

ELIGIBILITY:
Inclusion Criteria:

All adult patients (> 18yrs), ASA I-III, undergoing elective therapeutic/diagnostic Head & Neck surgeries under General Anaesthesiain the Minor OT complex and discharged on the same day will be included. The surgeries will include Head & Neck surgeries like DL scopies, laser surgeries, EUA, excision biopsies etc.

Exclusion Criteria:

1. Patients refusing to take part in study
2. Patients undergoing emergency surgeries
3. ASA IV patients, or high risk patients planned for admission
4. Admitted patients for minor OT procedure
5. Patients not getting the Information leaflet due to any reason (in 2nd half of study)
6. Patient and his attendant, both illiterate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2017-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sumitra G Bakshi, Principal Investigator — Professor, Department of Anesthesia, Critical Care and Pain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pre Intervention | Post Intervention
Started | 232 | 217
Completed | 232 | 196
Not Completed | 0 | 21
Not completed — Not received PIL in post PIL phase | 0 | 21

BASELINE CHARACTERISTICS:
Population: For primary endpoint -Total no of patients who underwent procedure under GA and the no of postponements in the minor OT in the given time frame was captured. All patients were not enrolled in the feedback process.
  For secondary endpoint - patients were enrolled after screening, consenting and feedback was collected from the them
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre Intervention | Post Intervention | Total
Number analyzed (Participants) | 232 | 196 | 428
Age, Customized [Count of Participants; unit: Participants]
  18-44 years | 57 | 37 | 94
  44-59 years | 79 | 74 | 153
  60 years and above | 84 | 68 | 152
  Data missing | 12 | 17 | 29
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 176 | 148 | 324
  Female | 36 | 34 | 70
  Data missing | 20 | 14 | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Education [Count of Participants; unit: Participants]
  Illiterate | 38 | 27 | 65
  School | 71 | 74 | 145
  Graduate | 46 | 31 | 77
  Post Graduate | 18 | 11 | 29
  Data missing | 59 | 53 | 112
Person filling form [Count of Participants; unit: Participants]
  Patient | 53 | 43 | 96
  Attendent | 116 | 73 | 189
  Data missing | 63 | 80 | 143

OUTCOME MEASURES:

1. Primary Outcome: Number of Cases Postponed Due to Lack of Information to Patients in the Pre-operative Period
Description: Cases postponed will be recorded and those caused due to lack of information of basic instruction to be followed prior to a procedure under GA will be recorded as an event.
Time Frame: On scheduled minor operative procedure day
Population: Number participants analysed depends upon the number of patients visited to the minor ot complex during assigned time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre Intervention | Post Intervention
Number analyzed (Participants) | 472 | 573
Participants | 56 | 44

2. Secondary Outcome: Satisfaction About Information With Respect to Instructions to be Followed
Description: Patients satisfaction with respect to instruction to be followed with administration of GA will be captured on a five point Likert scale -(5-Excellent, 4-Very good, 3-Good, 2-Poor, 1-Very poor)
Time Frame: On scheduled minor operative procedure day
Measure: Count of Participants; unit: Participants
Arm/Group | Pre Intervention | Post Intervention
Number analyzed (Participants) | 232 | 196
Participants
  Info about instructions to follow before surgery: Excellent | 41 | 45
  Info about instructions to follow before surgery: Very good | 60 | 82
  Info about instructions to follow before surgery: Good | 100 | 61
  Info about instructions to follow before surgery: Poor | 4 | 1
  Info about instructions to follow before surgery: Data missing | 27 | 7
  Info about instructions to follow after surgery: Excellent | 38 | 54
  Info about instructions to follow after surgery: Very good | 62 | 65
  Info about instructions to follow after surgery: Good | 86 | 60
  Info about instructions to follow after surgery: Poor | 6 | 1
  Info about instructions to follow after surgery: Data missing | 40 | 16

ADVERSE EVENTS:
Time Frame: 24 hours
Description: No adverse events noted
Groups:
- Pre Intervention: prior to introduction of patient information leaflet
- Post Intervention: after introduction of patient information leaflet
Arm/Group | Pre Intervention | Post Intervention
All-Cause Mortality (participants affected / at risk) | 0/232 | 0/196
Serious Adverse Events (participants affected / at risk) | 0/232 | 0/196
Other Adverse Events (participants affected / at risk) | 0/232 | 0/196
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre Intervention (N=232) | Post Intervention (N=196)
No adverse events noted (Social circumstances) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
1. Disease specific information not incorporated
2. Did not assess the patient anxiety regarding the PIL

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2016-11-05): https://cdn.clinicaltrials.gov/large-docs/40/NCT03011840/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-08-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT03011840/Prot_SAP_001.pdf